CLINICAL TRIAL: NCT06897202
Title: A Phase 2b, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Once-Weekly MET097 in Adults With Obesity or Overweight, and Type 2 Diabetes Mellitus (VESPER-2)
Brief Title: A Study to Evaluate the Efficacy and Safety of Once-Weekly MET097 in Adults With Obesity or Overweight and T2DM
Acronym: VESPER-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Metsera, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MET097-24-202
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Obesity in Diabetes; Type 2 Diabetes Mellitus (T2DM)
Keywords: GLP-1; Metsera; T2DM; Obesity; Overweight; Weight Loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MET097 Active with titration (Experimental)
  Interventions: Drug: MET097 Injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MET097 Active without titration (Experimental)
  Interventions: Drug: MET097 Injection

INTERVENTIONS:
Drug: MET097 Injection — MET097 is an ultra-long-acting, fully-biased analog of human GLP-1.
  Arms: MET097 Active with titration; MET097 Active without titration
Drug: Placebo — Sterile 0.9% (w/v) saline will be used as placebo treatment during the study.
  Arms: Placebo

SUMMARY:
This study is designed to test how well once-weekly MET097 (an ultra-long-acting GLP-1 receptor agonist) works to treat adults with obesity or overweight and type 2 diabetes mellitus (T2DM) compared to placebo. MET097 or placebo will be administered to individuals via subcutaneous injection once weekly for 28 weeks. If an individual is randomly assigned to MET097 they will receive one of four different dose regimens.

DETAILED DESCRIPTION:
This is a 28-week, multi-center, randomized, double-blind, placebo-controlled, parallel-group study to investigate the efficacy, safety, and tolerability of four different once-weekly MET097 dosing regimens vs. placebo for body weight loss in adults (18-75 years of age) with obesity or overweight (body mass index [BMI] ≥27 to ≤50 kg/m2) and T2DM . After completing 28 weeks of study treatment, all participants will be followed for approximately 11 weeks after administration of the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥27.0 kg/m2 to ≤50.0 kg/m2 at screening
* Type 2 diabetes mellitus (*T2DM) for at least 3 months before screening
* Glycated hemoglobin (HbA1c) value between ≥7.0% (53.0 mmol/mol) and ≤10.5% (91.3 mmol/mol) at Screening and treated with stable therapy for at least 30 days prior to Screening/Visit 1 (diet and exercise alone or in combination with metformin monotherapy and/or SGLT-2)
* Stable body weight (increase or decrease ≤5 kg) within 3 months prior to screening

Exclusion Criteria:

* Female who is lactating or who is pregnant
* Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2
* Fasting triglycerides ≥ 5.6 mmol/L (≥500 mg/dL)
* Poorly controlled hypertension
* History of stroke
* Significant cardiovascular disease including but not limited to unstable angina or valvular heart disease or has a history of myocardial infarction, coronary artery bypass graft, percutaneous coronary artery re-vascularization, or congestive heart failure
* Diagnosis of Type 1 diabetes (history of ketoacidosis, hyperosmolar state/coma, or any other types of diabetes except T2DM)
* History of acute or chronic pancreatitis
* Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder within the last 2 years
* Relevant surgical history including all bariatric or weight loss surgeries
* SGLT2 inhibitors and/or metformin
* Had 1 or more episodes of hypoglycemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in body weight at Week 28 (Day 197) | Baseline (Week 0) through Week 28 (Day 197)

SECONDARY OUTCOMES:
Weight reduction (weight loss) from baseline that is ≥ 5% | Baseline (Week 0) through Week 28 (Day 197)
Weight reduction (weight loss) from baseline that is ≥ 10% | Baseline (Week 0) through Week 28 (Day 197)
Weight reduction (weight loss) from baseline that is ≥ 15% | Baseline (Week 0) through Week 28 (Day 197)
Change in glycated hemoglobin A1c (HbA1c) | Baseline (Week 0) through Week 28 (Day 197)
Change from baseline in fasting plasma glucose (FPG) | Baseline (Week 0) through Week 28 (Day 197)
Change from baseline in fasting serum insulin | Baseline (Week 0) through Week 28 (Day 197)
Change from baseline in C-peptide | Baseline (Week 0) through Week 28 (Day 197)
Occurrence of HbA1c <7.0% (53.0 mmol/mol) | Baseline (Week 0) through Week 28 (Day 197)
Occurrence of HbA1c ≤6.5% (47.5 mmol/mol) | Baseline (Week 0) through Week 28 (Day 197)
Occurrence of HbA1c <5.7% (38.8 mmol/mol) | Baseline (Week 0) through Week 28 (Day 197)
Occurrence of treatment-emergent adverse events (TEAEs) | Baseline (Week 0) through Week 39 (Day 274)
  Treatment emergent adverse events include adverse events of clinical interest as well as abnormal clinical significant physical exams, laboratory findings, and 12-lead ECG measurements that meet the definition for an AE.
Occurrence of hypoglycemia according to American Diabetes Association classifications [ADA 2024] | Baseline (Week 0) through Week 39 (Day 274)
Occurrence of anti-drug antibodies | Baseline (Week 0) through Week 39 (Day 274)
Change from baseline in serum albumin | Baseline (Week 0) through Week 39 (Day 274)
Change from baseline in transthyretin [pre-albumin] | Baseline (Week 0) through Week 39 (Day 274)
Change from baseline in high-sensitivity C-reactive Protein [hsCRP] | Baseline (Week 0) through Week 39 (Day 274)
Characterize the minimum observed concentration (Cmin) | Baseline (Week 0) through Week 39 (Day 274)
Characterize the maximum observed concentration (Cmax) | Baseline (Week 0) through Week 39 (Day 274)
Characterize the area under the concentration versus time curve (AUC) | Baseline (Week 0) through Week 39 (Day 274)
Characterize the time to maximum concentration (Tmax) | Baseline (Week 0) through Week 39 (Day 274)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - Research Site US-97202-001012, Chula Vista, California
  - Research Site US-97202-001019, Los Alamitos, California
  - Research Site US-97202-001021, Los Angeles, California
  - Research Site US-97202-001007, Riverside, California
  - Research Site US-97202-001024, Bradenton, Florida
  - Research Site 097202-001001, Hollywood, Florida
  - Research Site 097202-001003, Tampa, Florida
  - Research Site 097202-001002, Decatur, Georgia
  - Research Site US-97202-001009, Riverdale, Georgia
  - Research Site 097202-001005, Savannah, Georgia
  - Research Site US-97202-001017, Morton, Illinois
  - Research Site US-97202-001022, Naperville, Illinois
  - Research Site US-97202-001008, Kansas City, Kansas
  - Research Site US-97202-001015, Columbia, Maryland
  - Research Site US-97202-001006, Gaithersburg, Maryland
  - Research Site US-97202-001004, Marlton, New Jersey
  - Research Site US-97202-001016, Charlotte, North Carolina
  - Research Site 097202-001010, Cincinnati, Ohio
  - Research Site US-97202-001023, Plano, Texas
  - Research Site US-97202-001013, Sherman, Texas